CLINICAL TRIAL: NCT00618657
Title: A Phase II Study of Breast Cancer Treatment Using Weekly Carboplatin+Nab-paclitaxel, Plus Trastuzumab (HER2+) or Bevacizumab (HER2-) in the Neoadjuvant Setting
Brief Title: Carboplatin+Nab-paclitaxel, Plus Trastuzumab (HER2+) or Bevacizumab (HER2-) in the Neoadjuvant Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rita Sanghvi, Mehta, HS Clinical Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20076084; UCI 07-61 (Other: CFCCC); NCI-2010-00155 (Other: NCI Clinical Trials Reporting Program (CTRP)); R01CA127927 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; HER2-positive Breast Cancer; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: pre-operative; neo-adjuvant; triple negative; HER2 positive; hormone receptor positive; breast; Carboplatin; Nab-paclitaxel; Trastuzumab; Bevacizumab; Inflammatory
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Taxes; 130-nm albumin-bound paclitaxel; Bevacizumab; Trastuzumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (HER-2 positive) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes, carboplatin IV over 60 minutes, and trastuzumab IV over 90 minutes , then weekly over 30-60 minutes. Treatment repeats every week for 12 weeks in the absence of disease progression or unacceptable toxicity. In both arms, beginning 21-40 days later, patients undergo surgery.
  Interventions: Drug: Carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: trastuzumab; Procedure: magnetic resonance imaging; Procedure: therapeutic conventional surgery
- Arm II (HER-2 negative) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation and carboplatin as in Arm I. Patients also receive bevacizumab IV over 90 or 60 or 30 minutes once every two weeks for 5 doses in the absence of disease progression or unacceptable toxicity. In both arms, beginning 21-40 days later, patients undergo surgery.
  Interventions: Drug: Carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: bevacizumab; Procedure: magnetic resonance imaging; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Carboplatin Hexal; Carboplatino; CBDCA
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: Albumin-Stabilized Nanoparticle Paclitaxel; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel; Nanoparticle Paclitaxel
Drug: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; recombinant humanized anti-VEGF monoclonal antibody; rhuMAb VEGF
  Arms: Arm II (HER-2 negative)
Drug: trastuzumab — Given IV
  Other Names: anti-c-erB-2; MOAB HER2; monoclonal antibody c-erb-2; monoclonal antibody HER2; rhuMAb HER2
  Arms: Arm I (HER-2 positive)
Procedure: magnetic resonance imaging — Optional correlative studies
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: therapeutic conventional surgery — Post-chemotherapy surgery for patients with a response or stable disease must take place no sooner than 21 days after last dose of Herceptin; and 40 days after last dose of bevacizumab to allow for normalization of blood counts

SUMMARY:
This phase II is studying the side effects and how well carboplatin and paclitaxel albumin-stabilized nanoparticle formulation when together with bevacizumab or trastuzumab before surgery works in treating patients with stage I-III breast cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab and trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving more than one drug (combination chemotherapy) and monoclonal antibody therapy together before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate 2 year progression-free survival in patients with breast cancer more than 1 cm and/or lymph node positive breast cancer treated with weekly Carboplatin/Nab-Paclitaxel (with trastuzumab in patients with HER2+ disease, and with bevacizumab in HER2-).

II. To measure clinical response rates in patients treated in the neoadjuvant setting.

III. To measure the microscopic pathological response rate of this regimen in patients treated in the neoadjuvant setting.

IV. To measure the toxicity and delivered dose intensity of this regimen. V. To assess the association between microscopic pathologic complete response and clinical complete response at the primary tumor site in these patients.

VI. To measure the outcome of patients treated with doxorubicin and cyclophosphamide with patients not treated with doxorubicin and cyclophosphamide.

SECONDARY OBJECTIVES:

I. Develop quantitative analysis methods to obtain pre-treatment tumor characteristic morphological, enhancement kinetic, and Choline metabolic parameters in breast cancer. Select an optimal set of features using the logistic regression analysis and the Artificial Neural Network (ANN) to predict pathologic complete remission (pCR) in HER-2 positive and negative arm.

II. Investigate whether the early response patterns, analyzed using the percent tumor size changes, or changes in other lesion characteristic parameters, can be used to predict pathologic complete remission (pCR) in HER-2 positive and negative arm.

III. Investigate whether combining the pre-treatment tumor characteristic parameters, and the early response pattern during the treatment course, can achieve a higher "area under the receiver operating characteristic (ROC) curve" (AUC) in prediction of pCR than those based on pre-treatment MRI characteristics or tumor response patterns alone.

OUTLINE: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and carboplatin IV over 60 minutes once weekly for 12 weeks. Patients with HER2-positive disease receive trastuzumab IV over 30-90 minutes once weekly for 12 weeks and patients with HER2-negative disease receive bevacizumab IV over 30-90 minutes once every two weeks for 5 doses. Treatment continues in the absence of disease progression or unacceptable toxicity. Beginning 21-40 days later, patients undergo surgery.

After completion of study treatment, patients are followed for 5 years.

ELIGIBILITY:
* Patients must be women with a histologically confirmed diagnosis of breast cancer that is more than 1 cm and or lymph node positive
* Physical examination, and scans needed for tumor assessment must be performed within 90 days prior to registration
* Patients with the clinical diagnosis of congestive heart failure or angina pectoris are NOT eligible
* Serum creatinine within normal limits within 90 days prior to registration
* Bilirubin within normal limits within 90 days prior to registration
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 2 x the institutional upper limit of normal within 90 days prior to registration
* Absolute neutrophil count (ANC) of >= 1,500/microliters within 90 days prior to registration
* Platelet count of >= 100,000/microliters within 90 days prior to registration
* Patients must have a performance status of 0-2 by Zubrod criteria
* Pregnant or nursing women may not participate; women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method; pregnancy test required for women of childbearing potential
* In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines; if day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-02; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mehta, M.D., Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative)
Started | 42 | 85
Completed | 42 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative) | Total
Number analyzed (Participants) | 42 | 85 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 80 | 118
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 85 | 127
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 36 | 50
  Not Hispanic or Latino | 28 | 49 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 18 | 53 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 14 | 22
Region of Enrollment [Number; unit: participants]
  United States | 42 | 85 | 127

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression is defined as a new lesion or a greater than or equal to 25% increase in the product of the largest perpendicular diameters of any one lesion on clinical exam or by ultrasound (U/S) or MRI. Analyzed using the Kaplan-Meier method. Cox proportional-hazards analysis will be used to derive the hazard ratio and 95% confidence interval between the two treatment arms, adjusted for clinical and demographic variables.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Groups:
- Arm I (HER-2 Positive): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes, carboplatin IV over 60 minutes, and trastuzumab IV over 90 minutes , then weekly over 30-60 minutes. Treatment repeats every week for 12 weeks in the absence of disease progression or unacceptable toxicity. In both arms, beginning 21-40 days later, patients undergo surgery.
  Carboplatin: Given IV paclitaxel albumin-stabilized nanoparticle formulation: Given IV trastuzumab: Given IV magnetic resonance imaging: Optional correlative studies therapeutic conventional surgery: Post-chemotherapy surgery for patients with a response or stable disease must take place no sooner than 21 days after last dose of Herceptin; and 40 days after last dose of bevacizumab to allow for normalization of blood counts
- Arm II (HER-2 Negative): Patients receive paclitaxel albumin-stabilized nanoparticle formulation and carboplatin as in Arm I. Patients also receive bevacizumab IV over 90 or 60 or 30 minutes once every two weeks for 5 doses in the absence of disease progression or unacceptable toxicity. In both arms, beginning 21-40 days later, patients undergo surgery.
  Carboplatin: Given IV paclitaxel albumin-stabilized nanoparticle formulation: Given IV bevacizumab: Given IV magnetic resonance imaging: Optional correlative studies therapeutic conventional surgery: Post-chemotherapy surgery for patients with a response or stable disease must take place no sooner than 21 days after last dose of Herceptin; and 40 days after last dose of bevacizumab to allow for normalization of blood counts
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative)
Number analyzed (Participants) | 42 | 85
percentage of participants | 95 | 93
Statistical Analysis 1: Comparison: Arm I (HER-2 Positive); Test type: Other; Standard Error = 0.03
Statistical Analysis 2: Comparison: Arm II (HER-2 Negative); Test type: Other; Standard Error = 0.03

2. Secondary Outcome: Clinical Complete Response in the Neoadjuvant Setting
Description: Defined as normal breast on physical exam. No mass, no thickening, no erythema, no peau d'orange. The 95% confidence interval (CI) will be computed.
Time Frame: Up to 5 years
Population: Clinical complete response data was not collected.
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With no Evidence of Microscopic pCR in the Neoadjuvant Setting
Description: Defined as no evidence of microscopic invasive tumor at the primary tumor site in the surgical specimen. The 95% CI will be computed.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative)
Number analyzed (Participants) | 42 | 85
Participants | 21 | 15

4. Secondary Outcome: Number of Participants With Toxicity of the Combinations in HER2 Positive and HER2 Negative Breast Cancer Assessed Using the National Cancer Institute (NCI) Common Toxicity Criteria Version 3.0
Description: The frequency of toxicities will be recorded.
Time Frame: Up to 5 years
Population: See adverse events section for complete report of adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative)
Number analyzed (Participants) | 42 | 85
Participants | 19 | 50

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Toxicity was graded according to National Cancer Institute Common Terminology Criteria of Adverse Events, version 5.0. Safety was assessed through adverse event monitoring, physical examinations, vital signs and clinical laboratory tests before each dosing.
Arm/Group | Arm I (HER-2 Positive) | Arm II (HER-2 Negative)
All-Cause Mortality (participants affected / at risk) | 5/42 | 11/85
Serious Adverse Events (participants affected / at risk) | 2/42 | 1/85
Other Adverse Events (participants affected / at risk) | 19/42 | 50/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (HER-2 Positive) (N=42) | Arm II (HER-2 Negative) (N=85)
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (HER-2 Positive) (N=42) | Arm II (HER-2 Negative) (N=85)
Neutropenia (Blood and lymphatic system disorders) | 14 | 29
Anemia (Blood and lymphatic system disorders) | 8 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6
Mucositis (Gastrointestinal disorders) | 1 | 3
Urinary Tract Infection (Renal and urinary disorders) | 2 | 9
Diarrhea (Gastrointestinal disorders) | 3 | 2
Peripheral Neuropathy (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
Nausea (General disorders) | 4 | 6
Rhinitis (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Amenorrhea (Reproductive system and breast disorders) | 0 | 1
Carboplatin Allergic Reaction (Product Issues) | 0 | 3
Vaginal Infection (Reproductive system and breast disorders) | 0 | 1
Hypertension (Blood and lymphatic system disorders) | 0 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Biliary Tract Infection (Gastrointestinal disorders) | 1 | 0
Epistaxis (General disorders) | 0 | 2
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Hot Flashes (General disorders) | 0 | 1
Tooth Infection (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nonhealing Would (Injury, poisoning and procedural complications) | 0 | 1
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT00618657/Prot_SAP_000.pdf